CLINICAL TRIAL: NCT05052489
Title: Establishment of a Prospective Cohort of Children With Diarrhoeal Disease Registry and Clinical Observation Study
Brief Title: Registry and Clinical Observation of Children With Diarrhoeal Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Mizu Jiang, Chief physician, professor, doctoral supervisor, secretary of gastroenterology group, pediatrics branch of Chinese medical association, pediatric gastroenterologist, Zhejiang University
Other Study IDs: MJiang-001
Record Dates: First submitted 2021-07-21; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Diarrhea
Keywords: probiotics; children
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: registy — Children with diarrhea were registered in the hospital. Baseline information of the children was recorded and followed up to observe the distribution of disease types, clinical manifestations, treatment plans and clinical outcomes

SUMMARY:
This Study based on the actual clinical diagnosis and treatment of data, evaluate the clinical characteristics of children with diarrhea Therapeutic effect and security, and establish the platform to childhood diarrhea registration, long-term accumulation of clinical data, develop the clinical characteristics and therapeutic effect of childhood diarrhea, safety monitoring data, and provide reliable data support for the clinical application.

DETAILED DESCRIPTION:
To evaluate the causes, clinical manifestations, treatment plans and clinical outcomes of diarrhoeal disease in children in a real diagnosis and treatment setting。 Evaluate the effect of different treatment schemes in actual clinical application,the clinical use of nutrition-supported zinc in oral rehydration fluids,the influencing factors of clinical efficacy, including the demographic characteristics and clinical characteristics of the children, as well as drug combination regimens, etc. To evaluate the clinical use of antibiotics,the clinical effects of different probiotics in the treatment of diarrhoeal disease in children,the effectiveness, safety and economy of the dose course of the clinical application of Clostridium butyricum bivariate living agents, the medical costs and resource consumption of treatment for diarrhoeal diseases in children.

ELIGIBILITY:
Inclusion Criteria:

* Under the age of 18

  * Children diagnosed with diarrhea, including:

    1. Acute diarrhea: infectious, such as viral bacteria, and non-infectious, such as improper diet and climate factors
    2. Persistent chronic diarrhea:

Including the following diseases:

1. Food allergy, food intolerance, indigestion, etc.;
2. Inflammatory bowel disease (IBD);
3. Diarrhoeal irritable bowel syndrome;
4. Antibiotic associated diarrhea (AAD);
5. Others: chronic hepatitis associated diarrhea, metabolic diseases associated diarrhea (such as diabetes mellitus with diarrhea), pancreatic exocrine dysfunction (cystic fibrosis), etc 3. Volunteered to participate in this study and signed the informed consent or the guardian signed the informed consent

Exclusion Criteria:

1. Class A infectious diseases associated with diarrhoea (cholera, plague)
2. Children with congenital heart disease, immune deficiency, malformation of digestive tract, or with severe dysfunction of heart, lung, liver and kidney。
3. Children receiving long-term immunosuppressive therapy (except children with IBD)。
4. Children with gastrointestinal surgery and tumor;
5. In addition to the above, the researchers determined that there were other children who were not suitable to participate in the study。

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Acute diarrhea: infectious, such as viral bacteria, and non-infectious, such as improper diet and climate factors
  2. Persistent chronic diarrhea,including: Food allergy, food intolerance, indigestion,Inflammatory bowel disease (IBD),Diarrhoeal irritable bowel syndrome,Antibiotic associated diarrhea (AAD),chronic hepatitis associated diarrhea, metabolic diseases associated diarrhea (such as diabetes mellitus with diarrhea), pancreatic exocrine dysfunction (cystic fibrosis), etc.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes of diarrhoeal disease in children | acute diarrhea up to 14 days；persistent diarrhea and chronic diarrhea up to 28 days
  symptom remission rate of children with diarrhoea

SECONDARY OUTCOMES:
Influencing factors of clinical outcomes | acute diarrhea up to 14 days；persistent diarrhea and chronic diarrhea up to 28 days
Direct medical costs | acute diarrhea up to 14 days；persistent diarrhea and chronic diarrhea up to 28 days
  including drugs, laboratory tests, treatment, emergency care, and other (all-cause) medical expenses
effectiveness of combined clostridium butyricum and bifidobacterium powders | acute diarrhea up to 14 days；persistent diarrhea and chronic diarrhea up to 28 days
  Change from baseline in stool consistency during the period of observation
safety evaluation | acute diarrhea up to 14 days；persistent diarrhea and chronic diarrhea up to 28 days
  The proportion of Adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Affiliated to Zhejiang University Medical College, Hangzhou, Zhejiang, China